CLINICAL TRIAL: NCT04914494
Title: Malignity Predictive Factors on Breast MRI With Ultrasound and Mammography Occult Lesions
Brief Title: Cancer Predictive Score on Breast MRI
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0379
Record Dates: First submitted 2021-06-02; First posted 2021-06-04 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer
Keywords: Women imaging; Diagnostic Imaging; Magnetic Resonance Imaging; Breast biopsy; Breast cancer detection; predictive factors; Radiology; Breast lesion diagnosis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sometimes, breast ultrasound and mammographic can't be diagnose suspsious lesions ( no substratum). So a MRI-guided breast biopsy is perfomed and disclosed ultimately benign lesions.

The aim of this retrospective study is to establish a predictive MRI score of occult breast lesions by mammography and ultrasound.

ELIGIBILITY:
Inclusion criteria:

* women aged 18 and more
* performed MRI-guided breast biopsy

Exclusion criteria:

- Not MRI-guided breast biopsy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged 18 to 50 years old
Sampling Method: Non-Probability Sample
Enrollment: 428 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with MRI characteristics of breast lesions | 1 day
  MRI characteristics of breast lesions :
  shape, contours, size, enhancement, perileeal edema, enhancement curve

SECONDARY OUTCOMES:
predictive score for the benignity of lesions seen on MRI | 1 day
  predictive score for the benignity of lesions seen on MRI (and not on mammography and ultrasound) with the criteria which will emerge after multivariate analysis and which will be weighted .
  score out of 10, with 3 to 5 criteria rated from 0 to 2. 10 would be in favor of benignity and 0 in favor of malignancy.

CONTACTS AND LOCATIONS:
Overall Officials: Patrice TAOUREL, MD.PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC